CLINICAL TRIAL: NCT02962362
Title: A Prospective Multi-center Data Collection to Assess the Exactech Guided Personalized Surgery eGPS® in Total Knee Arthroplasty
Brief Title: Study to Assess Exactech's Guided Personalized Surgery eGPS® in Total Knee Arthroplasty
Status: Terminated | Type: Observational
Why Stopped: Unable to complete enrollment of subjects.
Sponsor: Exactech (Industry)
Responsible Party: Sponsor
Other Study IDs: CR15-001
Record Dates: First submitted 2016-11-08; First posted 2016-11-11 (Estimated); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Study to collect outcomes data for patients who are undergoing an Exactech Optetrak® primary total knee replacement using the Exactech Guided Personalized Surgery (eGPS®) manufactured or distributed by (Exactech, Gainesville, Florida, USA).

DETAILED DESCRIPTION:
The purpose of this study is to collect patient outcomes data for patients who are undergoing an Exactech Optetrak® primary total knee replacement using the Exactech Guided Personalized Surgery (eGPS®) manufactured or distributed by (Exactech, Gainesville, Florida, USA). Patient outcomes data are important for assessing the post-market safety and effectiveness of orthopedic medical devices.

ELIGIBILITY:
Inclusion Criteria:

* Patient requires a primary Optetrak Logic Total Knee Arthroplasty
* Patient is skeletally mature with no obvious mechanical defect
* Patient is mentally capable of completing follow-up visits
* Patient is 18 years of age or greater at time of surgery
* Patient will be available for follow-up out to 2 years
* Patient has consented to participate in the clinical study

Exclusion Criteria:

* Patient has a mental or physical condition that may invalidate evaluation of the data
* Patient is a prisoner
* Surgery is contraindicated according to the applicable product package insert
* Patient has a local or systemic infection
* Patient has a known sensitivity to one or more of the materials in the knee replacement system to be used
* Patient is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: One hundred (100) subjects enrolled up to 4 sites. All subjects will be screened, enrolled and evaluated prospectively and be followed for up to two years. In the event a subject is enrolled and does not have surgery, additional patients may be screened and enrolled to reach the 100 subjects.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2016-08; Primary Completion 2019-07 (Actual); Study Completion 2021-11 (Actual)

PRIMARY OUTCOMES:
Hospital for Special Surgery knee score (HSS) | 24 Months
  total score, pain, function
Oxford Knee Score (OKS) | 24 Months
  function, pain
Knee Society Score (KSS) | 24 Months
  total score, pain, function
Knee injury and Osteoarthritis Outcome Score (KOOS) | 24 Months
  total score and subscales

CONTACTS AND LOCATIONS:
Locations (1):
- Exatech, Inc., Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No